CLINICAL TRIAL: NCT02186340
Title: Effects of Inspiratory Muscle Training on Breathing Pattern in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Daniel Langer, Dr Daniel Langer, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: S52852-2
Record Dates: First submitted 2014-07-03; First posted 2014-07-10 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Muscle Weakness Conditions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Inspiratory muscle training (Experimental)
  Interventions: Procedure: Inspiratory muscle training

INTERVENTIONS:
Procedure: Inspiratory muscle training

SUMMARY:
The improvement in inspiratory muscle function might result in beneficial changes in breathing pattern during whole body exercise. The hypothesis is the effect of inspiratory muscle training as an adjunct to a pulmonary rehabilitation program improves the breathing pattern during an incremental cycle exercise.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable COPD patients
* maximal inspiratory pressure <100% of the predicted normal value

Exclusion Criteria:

* Major comorbidities preventing successful participation in an 8 week exercise training intervention

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in breathing pattern during an incremental cycle exercise test | Baseline and 8 weeks follow-up
  At comparable levels of ventilation breathing frequency, inspiratory time (Ti), expiratory time (Te), total time of the respiratory cycle (Ttot), inspiratory duty cycle (Ti/Ttot), and inspiratory flow rates will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Rik PT Gosselink, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Charususin N, Gosselink R, McConnell A, Demeyer H, Topalovic M, Decramer M, Langer D. Inspiratory muscle training improves breathing pattern during exercise in COPD patients. Eur Respir J. 2016 Apr;47(4):1261-4. doi: 10.1183/13993003.01574-2015. Epub 2016 Feb 25. No abstract available. PMID 26917617